CLINICAL TRIAL: NCT00188214
Title: Dynamic CT Perfusion for Assessment of Lung Cancer Before and After Neoadjuvant Chemo-/ Radiotherapy
Brief Title: CT Perfusion Scans for Assessment of Lung Cancer Before and After Chemo +/- Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0420-CE
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: perfusion; CT; CAT; non-small; lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT perfusion scan (Other)
  Interventions: Procedure: contrast-enhanced dynamic CT perfusion study

INTERVENTIONS:
Procedure: contrast-enhanced dynamic CT perfusion study — contrast-enhanced dynamic CT perfusion study pre treatment and post treatment

SUMMARY:
Cancer of the lung is treated with surgery, radiation or chemotherapy, depending on the stage or extent of the disease. Some patients are treated with chemotherapy and/or radiation therapy before surgery to improve the results of surgery. After these treatments, we do not know whether the residual tumour tissue is still alive or dead, which is why some physicians feel that surgery is required to remove it.

This study is designed to assess if computed tomography (CT, CAT-scan) enhanced with intravenous contrast agent (dye) can characterize a lung cancer, and say whether it is alive or dead. The researchers hope that in the future such a contrast-enhanced CAT-scan will make surgery less often necessary or improve the results of chemotherapy and/or radiation given before surgery.

DETAILED DESCRIPTION:
The proposed study will be performed in patients with a proven lung cancer for whom induction therapy and subsequent surgical resection of any kind is planned. Kinetic analysis of dynamic contrast-enhanced CT will performed using the CT Perfusion 3 software (General Electric Medical Systems), yielding parameters characterizing tumor microvasculature in terms of the vascularity, or the blood volume (BV), the tumor perfusion or blood flow (BF), and the immaturity of the vascular wall, in terms of the microvascular permeability (permeability surface area, PS).

To test the assumption that dynamic CT-assessed tumor microvascular characteristics represent reliable, user-independent and reproducible parameters, microvascular values and parameter maps will be derived from two independent observers. To address the interobserver variability, each study will be analyzed by the PI and by a second researcher (blinded to the results of the PI). Kappa-statistics will be used to assess inter-rater concordance.

To test the hypothesis that the microvascular parameters obtained from dynamic contrast-enhanced CT predict the response to induction therapy, the parameters BV, BF and PS obtained prior to any treatment will be correlated with the histological result from the resected specimen (path CR or path non-CR). Spearman correlation will be used to compare non-parametric histology results with quantitative CT microvascular parameters.

To test the hypothesis that the microvascular parameters obtained from dynamic contrast-enhanced CT reflect the response to induction therapy, the parameters BV, BF and PS obtained after completion of induction treatment will be correlated with the histological result from the resected specimen (path CR or path non-CR). Spearman correlation will be used to compare non-parametric histology results with quantitative CT microvascular parameters.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of non-small cell lung cancer
* Patients who are scheduled for any neo-adjuvant treatment

Exclusion Criteria:

* Females who are known to be pregnant or nursing
* Patients with a history of adverse reaction to previous contrast agent administration
* Patients with known renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
-Analysis will be performed to yield quantitative, absolute estimates of blood volume, blood flow, and microvascular permeability. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi C Roberts, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada